CLINICAL TRIAL: NCT04914546
Title: A Single-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3819469
Brief Title: A Study of LY3819469 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 18075; J3L-MC-EZEA (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-06-01; First posted 2021-06-04 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3819469 (Part A) (Experimental): Single ascending doses of LY3819469 administered subcutaneously (SC).
  Interventions: Drug: LY3819469
- LY3819469 (Part B) (Experimental): Single doses of LY3819469 administered SC in Japanese Participants.
  Interventions: Drug: LY3819469
- Placebo (Part A) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo
- Placebo (Part B) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3819469 — Administered SC.
  Arms: LY3819469 (Part A); LY3819469 (Part B)
Drug: Placebo — Administered SC.
  Arms: Placebo (Part A); Placebo (Part B)

SUMMARY:
This is a 2-part study. In Part A, the main purpose is to evaluate the safety and tolerability of the study drug LY3819469 in healthy participants with high lipoprotein (a) [Lp(a)] levels. How the body processes the study drug and the effect of the study drug on blood Lp(a) levels will also be investigated. Part B will mainly evaluate the safety and tolerability of LY3819469 as well as how the body processes the study drug in Japanese participants. The study may last up to 53 and 29 weeks for each participant in Parts A and B, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Female participants must not be able to get pregnant and male participants must agree to adhere to contraception restrictions
* Have a body mass index (BMI) of 18.5 to 40.0 kilograms per square meter (kg/m²)
* For Part B, participants should be of first-generation Japanese origin

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days
* Are heavy alcohol drinkers or heavy cigarette smokers
* Have donated blood of more than 500 milliliters (mL) in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Week 49
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from Time Zero to Infinity (AUC[0-∞]) of LY3819469 | Predose through Day 15
  PK: AUC[0-∞] of LY3819469
PK: Maximum Observed Drug Concentration (Cmax) of LY3819469 | Predose through Day 15
  PK: Cmax of LY3819469
Pharmacodynamics (PD): Change From Baseline in Fasting Lp(a) | Baseline up to Week 49
  PD: Change From Baseline in Fasting Lp(a)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (4):
  - Altasciences Clinical Los Angeles, Inc, Cypress, California
  - Clinical Pharmacology of Miami, Miami, Florida
  - Qps-Mra, Llc, Miami, Florida
  - Endeavor Clinical Trials, San Antonio, Texas
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karp A, Jacobs M, Barris B, Labkowsky A, Frishman WH. Lipoprotein(a): A Review of Risk Factors, Measurements, and Novel Treatment Modalities. Cardiol Rev. 2025 Jul-Aug 01;33(4):352-358. doi: 10.1097/CRD.0000000000000667. Epub 2024 Feb 28. PMID 38415744
- [Derived] Nissen SE, Linnebjerg H, Shen X, Wolski K, Ma X, Lim S, Michael LF, Ruotolo G, Gribble G, Navar AM, Nicholls SJ. Lepodisiran, an Extended-Duration Short Interfering RNA Targeting Lipoprotein(a): A Randomized Dose-Ascending Clinical Trial. JAMA. 2023 Dec 5;330(21):2075-2083. doi: 10.1001/jama.2023.21835. PMID 37952254